CLINICAL TRIAL: NCT00195169
Title: Quality of Life After Myocardial Infarction: The Impact of Social Support
Brief Title: Quality of Life After Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Carla Boutin-Foster, Weill Cornell Medical College
Other Study IDs: 042677
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Social support
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to determine the association between social support and functional status after a myocardial infarct

DETAILED DESCRIPTION:
Primary objectives:

Our primary objective is to determine among patients hospitalized for a myocardial infarction, the impact of emotional support on functional outcomes at two years as measured by a valid measure of functional health, the SF-36.

Secondary Objectives:

Our secondary objectives are:

1. To determine the types of social support which are perceived as being most helpful to patients.
2. To determine whether women and minority patients have unique views on the types of support that are helpful.
3. To determine among patients admitted for myocardial infarction, the impact of social support on length of stay and hospital readmissions.

Hypothesis:

Our hypotheses are as follows:

1. Patients who are hospitalized for a myocardial infarction and who have high emotional support will have better long-term functional status compared to those patients who have low support.
2. Patients with high emotional support will be more likely to adhere to protocols such as taking their medications, keeping appointment, and enrolling in cardiac rehabilitation.
3. Patients with high emotional support will have lengths of hospitalization which are shorter than their estimated geometric mean as compared to patients who have low support.
4. The types of social support which are perceived as most helpful in disease management will be influenced by gender and ethnicity.

Long-term Objectives:

The long-term objective is to determine the mechanisms by which social support impacts on functional health and to utilize this data to develop future interventions that can be targeted toward a culturally and ethically diverse cohort of patients with coronary artery disease. Overall, the goal is to use this data to prevent functional disability and improve quality of life among patients with coronary artery disease.

ELIGIBILITY:
* Patients who have had a documented myocardial infarction by EKG and laboratory criteria will be eligible. The attending cardiologist of these patients will be approached. Once the attending cardiologist declares that a patient is clinically stable enough for participation, they will be approached, told about the study, and asked if they wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2001-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, Principal Investigator — Joan and Sanford I. Weill Medical College